CLINICAL TRIAL: NCT05153434
Title: A Phase 2, Single-Arm, Open-Label Study to Evaluate the Safety and Efficacy of ARD-101 in Patients With Prader-Willi Syndrome
Brief Title: A Study of Oral ARD-101 in Patients With Prader-Willi Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aardvark Therapeutics, Inc. (Industry)
Collaborators: Children's Hospital Colorado (Other); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AARD-203
Record Dates: First submitted 2021-11-30; First posted 2021-12-10 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-01

CONDITIONS: Prader-Willi Syndrome
MeSH Terms: conditions — Prader-Willi Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ARD-101 (Experimental): First week 400 mg of ARD-101 twice daily, second week 600 mg of ARD-101 twice daily, third week 800 mg of ARD-101 twice daily, fourth week 800 mg of ARD-101 twice daily.
  Interventions: Drug: ARD-101

INTERVENTIONS:
Drug: ARD-101 — Twice Daily, Oral Administration

SUMMARY:
A Phase 2, Single-Arm, Open-Label Study to Evaluate the Safety and Efficacy of ARD-101 in Patients with Prader-Willi Syndrome

DETAILED DESCRIPTION:
This is a Phase 2, open-label study to investigate the effects of ARD-101 in subjects with Prader-Willi Syndrome. The study will consist of a Screening Period (up to 28 days), a Treatment Period (28 days), and a Follow-up Period (End-of-Study Visit within 14 days after receiving the last dose of ARD-101). The screening procedures will be initiated upon completion of the informed consent process. Following completion of screening procedures and confirmation of eligibility, subjects will be enrolled to receive ARD-101 in an outpatient setting and will be instructed to visit the clinical center periodically for safety and efficacy assessments.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, 17-65 years of age
* Provide voluntary, written informed consent (parent(s) / legal guardian(s) of participant); provide voluntary, written assent (participants, as appropriate)
* PWS due to chromosome 15 micro-deletion, maternal uniparental disomy, or imprinting defect, confirmed by fluorescent in situ hybridization, chromosomal microarray, and/or methylation studies
* BMI ≥ 18.5 kg/m²
* A HQ-CT score ≥ 10
* If a subject has a diagnosis of type 2 diabetes, the following criteria must be met:

  1. Hemoglobin A1c (HbA1c) <7.5% not being managed with insulin. Patients taking glucagon-like peptide (GLP)-1 analogues (exenatide or liraglutide) must have been on stable dose for greater than 3 months.
  2. Fasting plasma glucose <140 mg/dL during the Screening Period
  3. No history of ketoacidosis or hyperosmolar coma
* Stable or well-controlled blood pressure (BP) and vital signs. Specifically: Vital signs after 5 minutes resting in seated position (feet flat on floor, back supported):

  1. 95 mmHg <systolic blood pressure (SBP) <160 mmHg
  2. 45 mmHg <diastolic blood pressure (DBP) <100 mmHg
  3. 40 bpm <heart rate (HR) <100 bpm
* Stable body weight for ~2 months (self or guardian-reported loss/gain within ± 10%) prior to enrollment
* Standard 12-lead ECG parameters after 10 minutes resting in supine position in the following ranges; 120 ms <PR <220 ms, QRS <120 ms, QTc ≤430 ms if male, ≤450 ms if female and normal ECG tracing unless the Investigator considers an ECG abnormality to be not clinically relevant.
* Parent or guardian is able to communicate well with the investigator, to understand and comply with the requirements of the study, and be able to understand and sign the written informed consent. Assent is to be provided for the patient who cannot consent for himself or herself
* Results of screening clinical laboratory tests [complete blood count (CBC) with differential and platelets and chemistry profile] and vital signs must be within normal range or, if outside of the normal range, must be accepted by the investigator and sponsor as not clinically significant
* Females of non-childbearing potential, defined as surgically sterile (status post hysterectomy, bilateral oophorectomy, or bilateral tubal ligation) or post-menopausal for at least 12 months (and confirmed with a screening FSH level in the post-menopausal lab range), do not require contraception during the study. This may also apply to subjects with documented hypogonadism with and without estrogen replacement therapy as per investigator judgement. All other females of child-bearing potential must agree to use contraception as outlined in the protocol
* Males with female partners of childbearing potential must agree to a double barrier method if they become sexually active during the study and for 90 days following the study.
* Patients previously treated with ARD-101 may be re-enrolled based on investigator decision and/if at least 3 months time has passed since the last dose.
* Patients must be on a stable dose of any allowed chronic concomitant medications while participating in the study, as described in protocol. This is defined as no changes in medication or dose for at least 30 days prior to Day 1 Stable concomitant usage (>3 months) of medications commonly used in PWS patients are allowed

Exclusion Criteria:

* Use of weight loss agents, including herbal medication, within 3 months prior to enrollment
* Diagnosis of schizophrenia, bipolar disorder, personality disorder, or other DSM-III disorders which the investigator believes will interfere significantly with study compliance
* A PHQ-9 score of ≥10
* Any suicidal ideation of type 4 or 5 on the C-SSRS
* Clinically significant illness in the 8 weeks prior to enrollment
* History of clinically significant bleeding disorders
* Current, clinically significant liver, renal, pulmonary, cardiac, oncologic, or gastrointestinal (GI) disease
* Diagnosis of type 1 diabetes mellitus or other active endocrine disorders (e.g., Cushing syndrome, or thyroid dysfunction except if on stable adequate thyroid or glucocorticoid replacement supplement)
* Liver disease or liver injury as indicated by abnormal liver function tests, SGOT (aspartate aminotransferase (AST)), alkaline phosphatase, or serum bilirubin (> 1.5 x upper limit of normal (ULN) for any of these tests) or history of hepatic cirrhosis
* History or presence of impaired renal function as indicated by clinically significantly abnormal creatinine, blood urea nitrogen (BUN), or urinary constituents (e.g., albuminuria) or moderate to severe renal dysfunction as defined by the Cockroft Gault equation (< 50 mL/min)
* Significant history of abuse of drugs within 1 year prior to enrollment or a positive Drugs of Abuse (DOA) test at screening
* History of alcohol abuse within 1 year prior to enrollment or currently drinks in excess of 21 units per week (3 servings or units/day)
* Caffeine consumption exceeding 6 cups of caffeinated tea/coffee (or equivalent) per day
* Participation in any clinical study with an investigational drug/device within 1 month prior to enrollment
* Serious adverse reaction or significant hypersensitivity to any drug
* Clinically significant blood loss or blood donation > 500 mL within 3 months prior to enrollment
* Inadequate venous access
* History of significant drug hypersensitivity or anaphylaxis
* Any condition that the investigator or primary physician believes may not be appropriate for participating the study

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-05-27 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2024-09-24 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAE) | Baseline to Day 28
  The incidence of treatment-emergent adverse events (TEAE) during the treatment period

SECONDARY OUTCOMES:
Efficacy Evaluation of Hyperphagia in Prader-Willi Syndrome | Baseline, Day 15, Day 28
  Quantitative evaluation of hyperphagia via the Hyperphagia Questionnaire for Clinical Trials (HQ-CT). Score will range from 0 (no hyperphagia behaviors) to 36 (most severe hyperphagia behaviors)
Effect on Weight | Baseline to Day 28
  Quantitative effect on weight during the course of treatment

OTHER OUTCOMES:
Effect on Anxiousness | Baseline to Day 28
  Evaluation of patient's anxiousness via the PWS anxiousness and distress questionnaire (PADQ) obtained at study visits.
The Change in Body Composition | Baseline to Day 28
  The change in body composition based on evaluation of dual-energy X-ray absorptiometry (DEXA) scans at the end of treatment compared to baseline
Effect on Psychiatric Status | Baseline to Day 28
  Effect on psychiatric status through screening presence of suicidal ideation and behavior in addition to screening for degree of depression via the Columbia-Suicide Severity Rating Scale (C-SSRS), as assessed by caregiver.
The Change in Body-Mass Index (BMI) | Baseline to Day 28
  The change in body-mass index (BMI) at the end of treatment from the baseline as well as 28 days after end of treatment
The Change in Waist Circumference | Baseline to Day 28
  The change in waist circumference at the end of treatment from the baseline as well as 14 days after end of treatment
Change in Patient Health | Baseline to Day 28
  Difference from Day 28 to baseline in patient health as assessed by Patient Health Questionnaire ((PHQ)-9 Questionnaires)
Change in Body Fat | Baseline to Day 28
  Estimation of body fat by bioelectric impedance analysis at the end of treatment compared to baseline
Change in GI Passage | Baseline to Day 28
  Change in GI passage time to explore potentially reduced constipation
Effect on Psychiatric Status | Baseline to Day 28
  Effect on psychiatric status as assessed by Patient Health Questionnaire ((PHQ)-9 Questionnaires)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Stanford University, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado

IPD SHARING:
Plan to Share IPD: No